CLINICAL TRIAL: NCT06301984
Title: Safety and Efficacy Evaluation of Insight GS Growing System in the Surgical Treatment of Early Onset Scoliosis (EOS)
Brief Title: Safety and Efficacy Evaluation of Insight GS Growing System
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EVEREST PESQUISA E DESENVOLVIMENTO LTDA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANDROMEDA_01_2023_V1
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Early Onset Scoliosis (EOS)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): In the initial assessment, data regarding the general health status will be collected and imaging exams (panoramic X-ray of the anteroposterior, lateral and traction spine, and X-ray of the right and left hands) and laboratory tests (blood count, coagulogram, dosage of sodium and potassium, urea and creatinine levels, AST and ALT, PCR, ESR, type I urine and urine culture) will be requested. During the preoperative consultation, measurements of the study variables will be obtained from the imaging exams), in addition to obtaining photographs of the patients. To install the Insight GS system, the surgical approach will be carried out according to the manufacturer's instructions for use, briefly described below. A posterior midline skin incision is made from the upper to the lower instrumented level. Subfascial exposure of the spine is performed, ensuring that the facet joint capsules are spared. Pedicle screws are inserted bilaterally at the cranial and caudal ends of the instrumentati
  Interventions: Device: Insight GS

INTERVENTIONS:
Device: Insight GS — The Andromeda Insight Growing System (Insight GS) is intended to treat severe, progressive multi-planar spinal deformities such as early-onset scoliosis while allowing for skeletal growth.
  The Andromeda Insight Growing System consists of blades, clamps and pedicle screws used to form a distinct spinal construct in growing children. The implanted blade is used to brace the spine during growth and minimize the progression of scoliosis. The components are implanted from a posterior approach and are made from Titanium alloy (Ti6AL-4V-ELI), and High Density Polyethylene (HDPE).

SUMMARY:
Premarket, interventional, single-arm clinical study, to evaluate the safety and efficacy of Insight GS Growing System in the surgical treatment of Early Onset Scoliosis (EOS). Also, to evaluate the difference in height of the spine and trunk, the success rate of the procedure, monitor adverse events and evaluate the satisfaction of the patient and care providers. The Andromeda Insight Growing System (Insight GS) is intended to treat severe, progressive multi-planar spinal deformities such as early-onset scoliosis while allowing for skeletal growth.

The Andromeda Insight Growing System consists of blades, clamps and pedicle screws used to form a distinct spinal construct in growing children. The implanted blade is used to brace the spine during growth and minimize the progression of scoliosis. The components are implanted from a posterior approach and are made from Titanium alloy (Ti6AL-4V-ELI), and High Density Polyethylene (HDPE).

Patients from 3 to 10 years of age, or who are still skeletally immature, who present early-onset scoliosis and who are considered as able to receive the surgical procedure with the Insight GS system, will be included in the study.

Patients will be screened in the outpatient setting of the study site. All participants who meet the eligibility criteria will be invited to participate in the study, which includes screening/pre-op, surgery to install the Insight GS system, and follow-up visits at 6 weeks, 2, 4, 6, 8, 10, 12,. 18 and 24 months for data collection, clinical evaluation, imaging, and monitoring of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* TCLE signed by parents
* Ages 3 to 10 years, or Risser 0, or Sanders 1,2,3 and 4
* Cobb angle bigger than 30°
* Thoracic spine height T1-T12 less than 22 centimeters
* Risk of thoracic insufficiency syndrome (TIS).

Exclusion Criteria:

* Need for fixation at occipital or cervical levels
* Risser sign greater than or equal to 1
* Sanders bigger than 4
* Previous spine surgery
* Medullary abnormalities
* Existence of malignant processes
* Local or systemic inflammations and infections, acute or chronic
* Allergy or intolerance to materials
* Non-reducible scoliosis
* Morbid obesity
* Insufficiency or absence of skin coverage

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Coronal Cobb angle change 24 months after installation of the Insight GS system. | 24 months after Insight GS System placement
  To determine the Cobb angle, a line will be used on the upper edge of the most inclined upper vertebra and on the lower edge of the most inclined lower vertebra, then the lines will be crossed and the measurement of the angle where they cross is the angle of Cobb. The measurement will be performed manually using conventional radiography and measuring the angle using the Cobb ruler.

SECONDARY OUTCOMES:
Number of Adverse event ocurrence assessed by clinical evaluation | 24 months after Insight GS System placement
  Adverse event monitoring
Changes in patient's trunk height assessed by T1 to T12 distance and the T1 to S1 distance on full-spine radiographs | 24 months after Insight GS System placement
  Spinal length will be assessed by measuring the T1 to T12 distance and the T1 to S1 distance on full-spine radiographs. The distance from T1 to T12 was measured as the length of a straight line joining the middle portion of the T1 vertebral end plate and the lower T12 vertebral end plate. Likewise, the distance T1 to S1 will be measured as the length of a direct line joining the middle portion of the upper end vertebral plate of T1 and the upper portion of the S1 vertebral end plate (8). The measurement will be carried out by a single operator, using conventional radiography and an analog ruler measured in centimeters.
Patients' pain assessed by Wong-Baker non-verbal facial scale | 24 months after Insight GS System placement
  To measure patients' pain, the Wong-Baker non-verbal facial scale will be used
Patient's satisfaction assessed by EOSQ-24 scale | 24 months after Insight GS System placement
  To assess the impact and satisfaction of treatment on caregivers or guardians, the Portuguese version of the 24-Item Early-Onset Scoliosis Questionnaire (EOSQ-24) scale will be used (10).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ortopédico AACD, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehdian H, Haddad S, Pasku D, Nasto LA. Mid-term results of a modified self-growing rod technique for the treatment of early-onset scoliosis. Bone Joint J. 2020 Nov;102-B(11):1560-1566. doi: 10.1302/0301-620X.102B11.BJJ-2020-0412.R3. PMID 33135451
- [Background] AlNouri M, Wada K, Kumagai G, Asari T, Nitobe Y, Morishima T, Uesato R, Aoki M, Ishibashi Y. Diseases and comorbidities associated with early-onset scoliosis: a retrospective multicenter analysis. Spine Deform. 2023 Mar;11(2):481-486. doi: 10.1007/s43390-022-00613-6. Epub 2022 Nov 16. PMID 36380109
- [Background] Ruiz G, Torres-Lugo NJ, Marrero-Ortiz P, Guzman H, Olivella G, Ramirez N. Early-onset scoliosis: a narrative review. EFORT Open Rev. 2022 Aug 4;7(8):599-610. doi: 10.1530/EOR-22-0040. PMID 35924646
- [Background] McCarthy RE, Luhmann S, Lenke L, McCullough FL. The Shilla growth guidance technique for early-onset spinal deformities at 2-year follow-up: a preliminary report. J Pediatr Orthop. 2014 Jan;34(1):1-7. doi: 10.1097/BPO.0b013e31829f92dc. PMID 23934092
- [Background] Sankar WN, Skaggs DL, Yazici M, Johnston CE 2nd, Shah SA, Javidan P, Kadakia RV, Day TF, Akbarnia BA. Lengthening of dual growing rods and the law of diminishing returns. Spine (Phila Pa 1976). 2011 May 1;36(10):806-9. doi: 10.1097/BRS.0b013e318214d78f. PMID 21336236
- [Background] Luhmann SJ, McCarthy RE. A Comparison of SHILLA GROWTH GUIDANCE SYSTEM and Growing Rods in the Treatment of Spinal Deformity in Children Less Than 10 Years of Age. J Pediatr Orthop. 2017 Dec;37(8):e567-e574. doi: 10.1097/BPO.0000000000000751. PMID 27043203
- [Background] undefined